CLINICAL TRIAL: NCT01446497
Title: Randomized, Multicenter, Open-label, Parallel Group Study to Evaluate Efficacy and Safety of Combigan(Brimonidine/Timolol) and 0.5% Timoptic(Timolol) Ophthalmic Solutions in Normal Tension Glaucoma Patients
Brief Title: Efficacy and Safety Study of Combigan and 0.5% Timoptic in Normal Tension Glaucoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1008-059-327; KHP01 (Registry Identifier: SNUH)
Record Dates: First submitted 2011-09-25; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Normal Tension Glaucoma
Keywords: Normal tension glaucoma; Antiglaucoma ophthalmic solution; Brimonidine; Timolol; Combination drugs
MeSH Terms: conditions — Low Tension Glaucoma | interventions — Brimonidine Tartrate; Brimonidine Tartrate, Timolol Maleate Drug Combination; Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Timolol (Active Comparator): non selective beta blocker, aqueous humor suppressant ophthalmic solution
  Interventions: Drug: Brimonidine/Timolol mixed combination
- Combigan (Timolol/Brimonidine) combination drug (Active Comparator): Brimonidine: alpha-2 agonist
  Interventions: Drug: Timolol

INTERVENTIONS:
Drug: Brimonidine/Timolol mixed combination — Twice per day, 1 drop at each time
  Other Names: Combigan
  Arms: Timolol
Drug: Timolol — Twice per day, 1 drop at each time
  Other Names: Timoptic XE
  Arms: Combigan (Timolol/Brimonidine) combination drug

SUMMARY:
Purpose To evaluate efficacy and safety of combigan(Brimonidine/Timolol) and 0.5% Timoptic (Timolol) ophthalmic solutions in normal tension glaucoma patients.

DETAILED DESCRIPTION:
* Normal tension glaucoma (NTG) is the major type of glaucoma in Korea. (over 90% of glaucoma type)
* Brimonidine (selective alpha 2 adrenergic agonist): neuroprotection effect by suppression of aqueous humor production and increasement of uveoscleral outflow
* Timolol (non selective beta blocker): suppression effect of aqueous humor production
* Combigan (fixed combination of brimonidine & timolol): more lowering effect of intraocular pressure and enhancing the compliance of glaucoma patients

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* baseline IOP under 22 mmHg,both anterior chamber angle > Grade 3~4 by Shaffer grading system

Exclusion Criteria:

* IOP over 22 mmHg by Goldmann applanation tonometer
* other types of glaucoma except open angle
* other IOP lowering treatment
* chronic or recurrent Hx. of ocular inflammation
* using contact lens
* any other ocular disease that could affect visual field examination (diabetic retinopathy, macular disease, uveitis, scleritis, optic neuritis, anterior ischemic optic neuropathy)
* intraocular or glaucoma surgery within 6 months
* Hx. of allergic reaction to timolol or brimonidine
* bronchial asthma
* moderate to severe chronic obstructive pulmonary disease
* heart failure
* 2~3 degree A-V block,
* MAO inhibitor use
* anti depressant use
* untreated pheochromocytoma
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in intraocular pressure at 12 weeks | 12 weeks after the initial treatment
  Intraocular pressure (IOP) check by Goldmann applanation tonometry with topical anesthetic eyedrop

CONTACTS AND LOCATIONS:
Overall Officials: Ki Ho Park, M.D, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea